CLINICAL TRIAL: NCT01998399
Title: Randomized Trial of Ticagrelor for Severe Community Acquired Pneumonia
Brief Title: Ticagrelor in Severe Community Acquired Pneumonia
Acronym: TCAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment, unable to meet recruitment goals
Sponsor: Gordon Bernard (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Gordon Bernard, Professor of Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 131908
Record Dates: First submitted 2013-11-15; First posted 2013-11-28 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Community Acquired Pneumonia, Severe
Keywords: CAP; Pneumonia; Intensive Care Unit; Mechanical Ventilation
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 180 mg loading dose followed by 90 mg BID for 90 days
  Interventions: Drug: Ticagrelor
- Placebo (Placebo Comparator): Placebo 180 mg loading dose followed by 90 mg BID for 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 180 mg loading dose followed by 90 mg BID for 90 days
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Placebo — Placebo 180 mg loading dose followed by 90 mg BID for 90 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the drug ticagrelor will be an effective treatment for patients with severe community acquired pneumonia. The primary objective is to reduce all-cause mortality in the ticagrelor group compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will have new "severe" CAP as defined by

a. New (within 72 hours of hospital admission) radiographic finding consistent with pneumonia and admission or planned admission to an ICU for: i. Mechanical Ventilation (invasive or non-invasive) OR ii. Vasopressors (dobutamine and phosphodiesterase are not considered vasopressors for this criteria) OR iii. ICU admission due to severe respiratory distress or arterial desaturation. b. At least two of the following; i. recent increase in dyspnea ii. increased sputum production iii. change of character of sputum iv. White Blood Cells > 12,000 or < 4,000 cells/mm3 or >10% bands v. Body temperature >38ºC or <36ºC (any route)

Exclusion Criteria:

1. More than 72 hours have passed since meeting required inclusion criteria.
2. Development of pneumonia after 72 hours of current hospitalization.
3. Underlying disease likely to cause mortality within 90 days of randomization.
4. A resident in a hospital, not nursing home, within 30 days prior to development of pneumonia.
5. Patients who are moribund (not expected to live for more than 48 hours).
6. No consent/inability to obtain consent from patient or surrogate.
7. Patient's physician is unwilling to have patient enter the study.
8. Age less than 50 years.
9. Pregnancy.
10. Breast feeding.
11. Underlying immunodeficiency (e.g. HIV, neutropenia, active hematologic malignancy, functional or anatomical asplenia and hypogammaglobulinemia).
12. Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she will receive all supportive care except for attempts at resuscitation from cardiac arrest).
13. Unable to receive or unlikely to absorb enteral study drug (e.g., patients with partial or complete mechanical bowel obstruction, intestinal ischemia, infarction, and short bowel syndrome).
14. Hepatic impairment

    a. Child Pugh score > 7 using data from outpatient setting
15. Conditions that increase the risk of bleeding, e.g.:

    1. Surgery or the likely need for surgery during study, or evidence of active bleeding postoperatively (ICU procedures such as line placement, tracheostomy and chest tubes are not to be considered for this exclusion);
    2. A history of severe head trauma requiring hospitalization or intra-cranial surgery within 3 months;
    3. Any history of intracerebral arteriovenous malformation, cerebral aneurysm, or mass lesions of the central nervous system, hemorrhagic stroke or intracranial hemorrhage, or congenital bleeding diathesis;
    4. Gastrointestinal bleeding within 6 weeks before the study unless a corrective procedure has been performed;
    5. Recent trauma considered to increase the risk of bleeding.
16. Chronic renal disease requiring renal replacement therapy.
17. Creatinine > 3 mg/dL.
18. Platelet count < 50,000 /mm3.
19. Use of a P2Y12 inhibitor within the 3 months prior to randomization or physician intent to initiate one of the CYP3A inhibitors, e.g. ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, atazanovir, saquinavir, nelfinavir, indinavir, or telithromycin.
20. Use of CYP3A inducers, e.g. rifampin, phenytoin, carbamazepine and phenobarbital.
21. Simvastatin or Lovastatin doses > 40 mg per day.
22. Digoxin use.
23. Receiving aspirin and physician and/or patient unwilling to reduce aspirin dose to <100 mg per day.
24. Daily Non-steroidal anti-inflammatory drugs (NSAID) use as an outpatient (other than Aspirin (ASA) as above).
25. Sick Sinus Syndrome, 2nd or 3rd degree heart block, bradycardia induced syncope - unless pacemaker in place.
26. Otherwise unsuitable for participation in the opinion of the investigator (i.e., homeless, non-compliant, etc.).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon R Bernard, MD, Principal Investigator — Vanderbilt University Medical Center; Jon D Truwit, MD, Principal Investigator — Medical College of Wisconsin
Locations (26):
- United States (26):
  - University of Arizona, Tucson, Arizona
  - University of Colorado, Colorado Springs, Colorado
  - Denver Health, Denver, Colorado
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Regions Hospital, Saint Paul, Minnesota
  - Moses Cone, Greensboro, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - Legacy Emanuel Medical Center, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor, Houston, Texas
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor | Placebo
Started | 12 | 13
Completed | 4 | 4
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 4 | 2
Not completed — Study stopped before dosing completed | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: death during 90 day study period
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
participants | 4 | 2
Statistical Analysis 1: Comparison: Ticagrelor vs Placebo; Total enrollment only 25 patients and the study was terminated early due to low enrollment. No further statistical analysis was done; Test type: Superiority or Other; p = 0.41, Chi-squared

2. Secondary Outcome: Shock Free Days
Description: Not requiring pressor support for hypotension
Time Frame: 15 days
Population: 2 participants from the Ticagrelor arm and 1 from the placebo arm died during the 15 day period
Measure: Mean (Full Range); unit: days
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
days | 12.58 [0 to 15] | 11.54 [0 to 15]

3. Secondary Outcome: Ventilator Free Days
Time Frame: 29 days
Population: 2 participants from each arm died during the 29 day period
Measure: Mean (Full Range); unit: days
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
days | 24.16 [16 to 29] | 22.3 [14 to 25]

4. Secondary Outcome: In-hospital Mortality
Description: Did the patient die during the hospitalization?
Time Frame: Throughout hospitalization (About 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 2 | 2

5. Secondary Outcome: Hospital Free Days
Description: Number of days the patient is not in the hospital
Time Frame: 29 days
Population: 2 participants from each group died during this time period
Measure: Mean (Full Range); unit: days
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
days | 14.16 [3 to 22] | 16.53 [2 to 25]

6. Secondary Outcome: Stroke
Description: Did the patient develop a stroke during the 90 day study?
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 1 | 0

7. Secondary Outcome: Stroke, Myocardial Infarct, Mortality
Description: number of participants that suffered stroke, myocardial infarct, mortality
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 5 | 2

8. Secondary Outcome: Myocardial Infarction
Description: Did the patient have a myocardial infarction during the 90 day study?
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 1 | 0

9. Other Pre Specified Outcome: Time to Initiation of Unassisted Breathing
Description: Only in patients on mechanical ventilation and assuming patient achieves 48 consecutive hours of unassisted breathing
Time Frame: 29 days
Population: 2 participants from each arm died during this period
Measure: Mean (Full Range); unit: hours
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 8 | 11
hours | 136.9 [49.5 to 310.5] | 173.19 [46.65 to 404.15]

10. Other Pre Specified Outcome: Need for Re-instituting Assisted or Mechanical Ventilation After Achieving 48 Consecutive Hours of Unassisted Breathing or Comfort Care Chosen (Withdrawal of Support)
Time Frame: 90 days
Population: only participants that required mechanical ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 8 | 11
Participants | 0 | 0

11. Other Pre Specified Outcome: Need for Dialysis
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 1 | 0

12. Other Pre Specified Outcome: ICU Length of Stay
Description: Includes ICU readmission if during same hospital stay
Time Frame: 29 days
Population: 2 participants from each arm died during this period
Measure: Mean (Full Range); unit: days
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
days | 8.33 [3 to 13] | 8.77 [2 to 22]

13. Other Pre Specified Outcome: Hospital Length of Stay
Description: In days
Time Frame: 29 days
Measure: Mean (Full Range); unit: days
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
days | 14.83 [4 to 26] | 12.46 [4 to 27]

14. Other Pre Specified Outcome: Discharge Disposition
Description: (Home, other facility, with or without assisted ventilation)
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Placebo
Number analyzed (Participants) | 12 | 13
Participants
  Home | 5 | 9
  Extended Care without Ventilator | 4 | 2
  Extended Care with Ventilator | 0 | 0
  In patient rehabilitation | 1 | 0
  Death prior to discharge | 2 | 2

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Ticagrelor | Placebo
Serious Adverse Events (participants affected / at risk) | 5/12 | 1/13
Other Adverse Events (participants affected / at risk) | 4/12 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=12) | Placebo (N=13)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Type II MI (Cardiac disorders) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Complicated Para-pneumonic Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis-Right Leg (Vascular disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=12) | Placebo (N=13)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukemoid Reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
dysgeusia (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Upper Gastrointestinal Bleed (Vascular disorders) | 1 (1) | 0 (0)
vaginal bleeding (Vascular disorders) | 1 (1) | 0 (0)
Hematoma on forearm (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No